CLINICAL TRIAL: NCT03256890
Title: Mindfulness-Based Blood Pressure Reduction: Stage 2a Randomized Controlled Trial
Brief Title: Mindfulness-Based Blood Pressure Reduction: Stage 2a RCT
Acronym: MB-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1412001171-3; 1UH2AT009145 (NIH)
Record Dates: First submitted 2017-08-03; First posted 2017-08-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Prehypertension
Keywords: mindfulness; blood pressure; hypertension; prehypertension; self regulation; Science of Behavior Change; attention control; self awareness; emotion regulation
MeSH Terms: conditions — Hypertension; Prehypertension; Self-Control; Emotional Regulation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will implement blinding of staff performing participant assessments and data analysts performing statistical analyses. The principal investigator will be blinded to group allocation, except for participants that he is involved with instructing in the MB-BP intervention (there are multiple instructors). The prinicipal investigator has no access to the master data file. Equipoise is emphasized for all staff who interact with participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB-BP Intervention (Experimental): MB-BP customizes Mindfulness-Based Stress Reduction (MBSR) to participants with hypertension. It consists of nine 2.5-hour weekly group sessions and a 7.5-hour one-day session. Content includes education on hypertension risk factors, hypertension health effects, and specific mindfulness modules focused on awareness of BP determinants such as diet, physical activity, anti-hypertensive medication adherence, alcohol consumption, and stress reactivity. Students learn a range of mindfulness skills including body scan exercises, meditation and yoga. Participants are given a home BP monitor. Participants with uncontrolled hypertension are offered to have their physicians notified; for those without a physician, we work to provide access within health insurance constraints.
  Interventions: Behavioral: MB-BP Intervention
- Enhanced Usual Care Control (Active Comparator): Control group participants receive an educational brochure from American Heart Association entitled "Understanding and Controlling Your High Blood Pressure Brochure" (product code 50-1639). Every participant is provided with a validated home blood pressure monitor (Omron, Model PB786N), that as an evidence-based approach to lower blood pressure, would be considered "enhanced usual care" at this time. All participants who have uncontrolled hypertension (blood pressure >140/90 mmHg) will be offered to have their physicians notified, if not already being overseen for uncontrolled hypertension. For participants with uncontrolled hypertension who do not have a physician, we work participants to provide access within constraints of their health insurance.
  Interventions: Other: Enhanced Usual Care Control

INTERVENTIONS:
Behavioral: MB-BP Intervention — MB-BP customizes Mindfulness-Based Stress Reduction (MBSR) to participants with hypertension. It consists of nine 2.5-hour weekly group sessions and a 7.5-hour one-day session. Content includes education on hypertension risk factors, hypertension health effects, and specific mindfulness modules focused on awareness of BP determinants such as diet, physical activity, anti-hypertensive medication adherence, alcohol consumption, and stress reactivity. Students learn a range of mindfulness skills including body scan exercises, meditation and yoga. Homework consists of practicing skills for ≥45 min/day, 6 days/week. Participants are given a home BP monitor. Participants with uncontrolled hypertension are offered to have their physicians notified, if not already overseen for uncontrolled hypertension; those without a physician are worked with to provide access within health insurance constraints.
  Arms: MB-BP Intervention
Other: Enhanced Usual Care Control — Control group participants receive an educational brochure from American Heart Association entitled "Understanding and Controlling Your High Blood Pressure Brochure" (product code 50-1639). Every participant is provided with a validated home blood pressure monitor (Omron, Model PB786N), that as an evidence-based approach to lower blood pressure, would be considered "enhanced usual care" at this time. All participants who have uncontrolled hypertension (blood pressure >140/90 mmHg) will be offered to have their physicians notified, if not already being overseen for uncontrolled hypertension. For participants with uncontrolled hypertension who do not have a physician, we work participants to provide access within constraints of their health insurance.
  Arms: Enhanced Usual Care Control

SUMMARY:
The primary aim is to evaluate impacts of a behavioral intervention called "Mindfulness-Based Blood Pressure Reduction" (MB-BP) vs. enhanced usual care control on systolic blood pressure at 6 months, via a randomized controlled trial.

DETAILED DESCRIPTION:
Effects of mindfulness interventions customized for prehypertensive/hypertensive patients are poorly understood. Until methodologically rigorous studies to evaluate customized interventions for hypertension are performed, it will be unknown whether the observed preliminary effects of general mindfulness interventions on blood pressure reduction could be much more effective with a tailored approach. Consequently, this study proposes to conduct a behavioral intervention study to evaluate whether Mindfulness-Based Stress Reduction (MBSR) customized to prehypertensive and hypertensive patients has the potential to provide clinically relevant reductions in blood pressure. This customized intervention is called Mindfulness-Based Blood Pressure Reduction (MB-BP). The study follows the NIH Stage Model for Behavioral Intervention Development, where targets likely proximally affected by the intervention are identified, that should also have effect on the longer-term outcomes (e.g. blood pressure, mortality). The selected targets, consistent with theoretical frameworks and early evidence how mindfulness interventions could influence mental and physical health outcomes, are measures of self-regulation including (1) attention control (specifically the Sustained Attention Response Task and Mindful Attention Awareness Scale), (2) emotion regulation (specifically the Pittsburgh Stress Battery and the Perceived Stress Scale), and (3) self-awareness (specifically the Heart Beat Detection Task and Multidimensional Assessment of Interoceptive Awareness). Based on the degree of target engagement, MB-BP can be further customized to better engage with the targets as needed.

Specific aims are as follows.

The primary aim is to evaluate impacts of MB-BP vs. enhanced usual care control on systolic blood pressure at 6 months. Follow-up time periods include 10 weeks and 6 months.

Secondary aims include evaluating impacts of MB-BP vs. enhanced usual care control on self-regulation mechanistic target engagement, including (1) attention control (specifically the Sustained Attention Response Task and Mindful Attention Awareness Scale), (2) emotion regulation (specifically the Pittsburgh Stress Battery and the Perceived Stress Scale), and (3) self-awareness (specifically the Heart Beat Detection Task and Multidimensional Assessment of Interoceptive Awareness). Further secondary aims include evaluating impacts of MB-BP vs. active control on medical regimen adherence, including (1) physical activity, (2) Dietary Approaches to Stop Hypertension (DASH)-consistent diet, (3) alcohol consumption, (4) body mass index, and (5) antihypertensive medication use and adherence. Secondary blood pressure outcomes include diastolic blood pressure.

This study is a randomized controlled trial, with blinding of staff performing participant assessments and data analysts performing statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension/prehypertension (≥120 mmHg systolic, ≥80 mmHg diastolic pressure or taking antihypertensive medication). Preference is given to recruiting uncontrolled hypertensives (≥140 mmHg systolic or ≥90 mmHg diastolic pressure)
* Able to speak, read, and write in English.
* All adults (≥18 years of age), genders and racial/ethnic groups are eligible to be included.

Exclusion Criteria:

* Current regular meditation practice (>once/week)
* Serious medical illness precluding regular class attendance
* Current substance abuse, suicidal ideation or eating disorder
* History of bipolar or psychotic disorders or self-injurious behaviors.

These participants are excluded because they may disrupt group participation, require additional or specialized treatment, or are already participating in practices similar to the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 6 month follow-up
  Directly assessed as mean of second and third blood pressure readings
Dietary Approaches to Stop Hypertension-consistent diet | 6 month follow-up
  Self-report via Willet Food Frequency Questionnaire

SECONDARY OUTCOMES:
Sustained Attention to Response Task (SART) | 6 month follow-up
  Behavioral measure of attention control
Mindful Attention Awareness Scale (MAAS) | 6 month follow-up
  Self-report measure of attention control and mindfulness
Pittsburgh Stress Battery | 6 month follow-up
  Behavioral measure of stress reactivity
Perceived Stress Scale | 6 month follow-up
  Self-report measure of perceived stress
Heartbeat Detection Task | 6 month follow-up
  Behavioral measure of self-awareness
Multidimensional Assessment of Interoceptive Awareness (MAIA) | 6 month follow-up
  Self-report measure of self-awareness
Physical Activity - self report | 6 month follow-up
  Self-report via International Physical Activity Questionnaire (IPAQ)
Physical Activity - step count | 6 month follow-up
  Directly assessed via FitBit step count
Alcohol consumption | 6 month follow-up
  Self-report via Willet Food Frequency Questionnaire
Body Mass Index | 6 month follow-up
  Directly assessed as weight (kg) per height (m) squared, using a validated stadiometer to assess height, and validated scale to measure weight.
Antihypertensive medication adherence | 6 month follow-up
  Directly assessed via eCAP medication adherence devices (Information Mediary Corp., Ottawa, ON, Canada). Please note that eCAP is the device name, and not an acronym.
Antihypertensive medication use | 6 month follow-up
  Directly assessed via medication bottle labels that participants bring to clinic assessments
Diastolic blood pressure | 6 month follow-up
  Directly assessed as mean of second and third readings

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Loucks, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Loucks EB, Kronish IM, Saadeh FB, Scarpaci MM, Proulx JA, Gutman R, Britton WB, Schuman-Olivier Z. Adapted Mindfulness Training for Interoception and Adherence to the DASH Diet: A Phase 2 Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2339243. doi: 10.1001/jamanetworkopen.2023.39243. PMID 37917063
- [Derived] Loucks EB, Kronish IM, Saadeh FB, Scarpaci MM, Proulx JA, Gutman R, Britton WB, Schuman-Olivier Z. Effects of Adapted Mindfulness Training on Interoception and Adherence to the Dietary Approaches to Stop Hypertension (DASH) Diet: The MB-BP Randomized Clinical Trial. medRxiv [Preprint]. 2023 May 15:2023.05.10.23289818. doi: 10.1101/2023.05.10.23289818. PMID 37292774
- [Derived] Loucks EB, Schuman-Olivier Z, Saadeh FB, Scarpaci MM, Nardi WR, Proulx JA, Gutman R, King J, Britton WB, Kronish IM. Effect of Adapted Mindfulness Training in Participants With Elevated Office Blood Pressure: The MB-BP Study: A Randomized Clinical Trial. J Am Heart Assoc. 2023 Jun 6;12(11):e028712. doi: 10.1161/JAHA.122.028712. Epub 2023 May 23. PMID 37218591
- [Derived] Polcari JJ, Cali RJ, Nephew BC, Lu S, Rashkovskii M, Wu J, Saadeh F, Loucks E, King JA. Effects of the Mindfulness-Based Blood Pressure Reduction (MB-BP) program on depression and neural structural connectivity. J Affect Disord. 2022 Aug 15;311:31-39. doi: 10.1016/j.jad.2022.05.059. Epub 2022 May 17. PMID 35594968